CLINICAL TRIAL: NCT01033071
Title: A Phase 3b, Double-Blind, Randomized, 12-Week Efficacy and Safety Study Comparing the TAK-491 Plus Chlorthalidone Fixed-Dose Combination vs Olmesartan Medoxomil-Hydrochlorothiazide in Subjects With Moderate to Severe Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil and Chlorthalidone Compared to Olmesartan Medoxomil and Hydrochlorothiazide in Participants With Moderate to Severe Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491CLD_303; U1111-1112-4298 (Registry Identifier: WHO)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-01

CONDITIONS: Essential Hypertension
Keywords: Hypertensive; Blood Pressure, High; Cardiovascular disease; Vascular Disease; Drug Therapy
MeSH Terms: conditions — Essential Hypertension; Hypertension; Cardiovascular Diseases; Vascular Diseases | interventions — azilsartan medoxomil; Chlorthalidone; Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD (Active Comparator)
  Interventions: Drug: Olmesartan medoxomil and hydrochlorothiazide

INTERVENTIONS:
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 20 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily and olmesartan and hydrochlorothiazide placebo-matching tablets, orally, once daily for up to 4 weeks.
  Participants will be force titrated at Week 4 to azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for the next 4 weeks.
  Participants will then be force titrated at Week 8 to azilsartan medoxomil 40 mg and chlorthalidone 25 mg combination tablets, orally, once daily for the next 4 weeks.
  Other Names: azilsartan medoxomil plus chlorthalidone; TAK-491CLD
  Arms: Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily and olmesartan and hydrochlorothiazide placebo-matching tablets, orally, once daily for up to 4 weeks.
  Participants will be force titrated at Week 4 to azilsartan medoxomil 80 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for the next 4 weeks.
  Participants will then be force titrated at Week 8 to azilsartan medoxomil 80 mg and chlorthalidone 25 mg combination tablets, orally, once daily for the next 4 weeks.
  Other Names: azilsartan medoxomil plus chlorthalidone; TAK-491CLD
  Arms: Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD
Drug: Olmesartan medoxomil and hydrochlorothiazide — Olmesartan medoxomil 20 mg and hydrochlorothiazide 12.5 mg combination tablets, orally, once daily and azilsartan medoxomil and chlorthalidone placebo-matching tablets, orally, once daily for up to 4 weeks.
  Participants will be force titrated at Week 4 to olmesartan medoxomil 40 mg and hydrochlorothiazide 12.5 mg combination tablets, orally, once daily for the next 4 weeks.
  Participants will then be force titrated at Week 8 to olmesartan medoxomil 40 mg and hydrochlorothiazide 25 mg combination tablets, orally, once daily for the next 4 weeks.
  Other Names: Benicar HCT®
  Arms: Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD

SUMMARY:
The purpose of this study is to compare the antihypertensive effect of azilsartan medoxomil plus chlorthalidone, once daily (QD), to olmesartan medoxomil plus hydrochlorothiazide in participants with moderate to severe hypertension.

DETAILED DESCRIPTION:
According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. Despite the availability of antihypertensive agents, hypertension remains inadequately controlled; only about one third of patients continue to maintain control successfully.

Treatment algorithms for essential hypertension commonly include thiazides or thiazide-like diuretics, either alone or as part of combination treatment. Chlorthalidone is a commercially available, orally administered thiazide-type diuretic agent.

TAK-491 (azilsartan medoxomil) is an angiotensin II receptor blocker developed by Takeda to treat participants with essential hypertension.

This study will compare the safety and tolerability of azilsartan medoxomil plus chlorthalidone (TAK-491CLD) fixed-dose combination to olmesartan medoxomil plus hydrochlorothiazide fixed-dose combination.

ELIGIBILITY:
Inclusion Criteria:

1. Has a mean sitting clinic systolic blood pressure greater than or equal to 160 and less than or equal to 190 mm Hg.
2. Females of childbearing potential who are sexually active agree to routinely use adequate contraception from Screening through 30 days after the last administered study drug dose.
3. Has clinical laboratory test results within the reference range for the testing laboratory or the investigator does not consider the results to be clinically significant.
4. Is willing to discontinue current antihypertensive medications on Day -21 or Day -28 if the participant is on amlodipine or chlorthalidone.

Exclusion Criteria:

1. Has a mean sitting clinic diastolic blood pressure greater than 119 mm Hg on Day -1.
2. Has a baseline 24-hour ambulatory blood pressure monitoring reading of insufficient quality.
3. Works a night (third) shift.
4. Has an upper arm circumference less than 24 cm or greater than 42 cm.
5. Has secondary hypertension of any etiology.
6. Has a recent history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
7. Has clinically significant cardiac conduction defects.
8. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
9. Has severe renal dysfunction or disease.
10. Has known or suspected unilateral or bilateral renal artery stenosis.
11. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug.
12. Has poorly-controlled diabetes mellitus at Screening.
13. Has hypokalemia or hyperkalemia.
14. Has an alanine aminotransferase or aspartate aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
15. Has any other known serious disease or condition that would compromise safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
16. Has known hypersensitivity to angiotensin II receptor blockers or thiazide-type diuretics or other sulfonamide-derived compounds.
17. Has a history of drug abuse or a history of alcohol abuse within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1071 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr VP Clinical Science, Study Director — Takeda
Locations (94):
- United States (84):
  - Gulf Shores, Alabama
  - Litchfield Park, Arizona
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Buena Park, California
  - Carmichael, California
  - Greenbrae, California
  - Irvine, California
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Spring Valley, California
  - Wildomar, California
  - Colorado Springs, Colorado
  - Milford, Connecticut
  - Waterbury, Connecticut
  - Newark, Delaware
  - Aventura, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Ocala, Florida
  - Plant City, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Haven, Florida
  - Dunwoody, Georgia
  - Roswell, Georgia
  - Suwanee, Georgia
  - Chicago, Illinois
  - Melrose Park, Illinois
  - Naperville, Illinois
  - Avon, Indiana
  - Indianapolis, Indiana
  - Valparaiso, Indiana
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Auburn, Maine
  - Brockton, Massachusetts
  - Hyannis, Massachusetts
  - West Yarmouth, Massachusetts
  - Ann Arbor, Michigan
  - City of Saint Peters, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Margate City, New Jersey
  - Wildwood Crest, New Jersey
  - Albuquerque, New Mexico
  - Glens Falls, New York
  - Boiling Springs, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Yukon, Oklahoma
  - Ashland, Oregon
  - Portland, Oregon
  - Bensalem, Pennsylvania
  - Feasterville, Pennsylvania
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Tipton, Pennsylvania
  - Cranston, Rhode Island
  - Cumberland, Rhode Island
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Beaumont, Texas
  - Dallas, Texas
  - Houston, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Magna, Utah
  - Manassas, Virginia
  - Lakewood, Washington
  - Port Orchard, Washington
  - Madison, Wisconsin
  - Menomonee Falls, Wisconsin
- Canada (10):
  - Abbotsford, British Columbia
  - Powell River, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - London, Ontario
  - Ottawa, Ontario
  - Sarnia, Ontario
  - Vaughan, Ontario
  - Whitby, Ontario
  - Woodstock, Ontario

REFERENCES:
- [Derived] Cushman WC, Bakris GL, White WB, Weber MA, Sica D, Roberts A, Lloyd E, Kupfer S. Azilsartan medoxomil plus chlorthalidone reduces blood pressure more effectively than olmesartan plus hydrochlorothiazide in stage 2 systolic hypertension. Hypertension. 2012 Aug;60(2):310-8. doi: 10.1161/HYPERTENSIONAHA.111.188284. Epub 2012 Jun 18. PMID 22710649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 130 investigative sites in Canada and the United States from 08 December 2009 to 04 November 2010.
Pre-assignment Details: Participants with essential hypertension were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD: Azilsartan medoxomil 20 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily and olmesartan and hydrochlorothiazide placebo-matching tablets, orally, once daily for up to 4 weeks.
  Participants will be force titrated at Week 4 to azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for the next 4 weeks.
  Participants will then be force titrated at Week 8 to azilsartan medoxomil 40 mg and chlorthalidone 25 mg combination tablets, orally, once daily for the next 4 weeks.
- Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD: Azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily and olmesartan and hydrochlorothiazide placebo-matching tablets, orally, once daily for up to 4 weeks.
  Participants will be force titrated at Week 4 to azilsartan medoxomil 80 mg and chlorthalidone 12.5 mg combination tablets, orally, once daily for the next 4 weeks.
  Participants will then be force titrated at Week 8 to azilsartan medoxomil 80 mg and chlorthalidone 25 mg combination tablets, orally, once daily for the next 4 weeks.
- Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD: Olmesartan medoxomil 20 mg and hydrochlorothiazide 12.5 mg combination tablets, orally, once daily and azilsartan medoxomil and chlorthalidone placebo-matching tablets, orally, once daily for up to 4 weeks.
  Participants will be force titrated at Week 4 to olmesartan medoxomil 40 mg and hydrochlorothiazide 12.5 mg combination tablets, orally, once daily for the next 4 weeks.
  Participants will then be force titrated at Week 8 to olmesartan medoxomil 40 mg and hydrochlorothiazide 25 mg combination tablets, orally, once daily for the next 4 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Started | 355 | 352 | 364
Completed | 300 | 275 | 317
Not Completed | 55 | 77 | 47
Not completed — Adverse Event | 28 | 51 | 26
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Lost to Follow-up | 4 | 5 | 5
Not completed — Withdrawal by Subject | 17 | 14 | 11
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Other | 6 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD | Total
Number analyzed (Participants) | 355 | 352 | 364 | 1071
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.49) | 56.7 (10.07) | 56.7 (10.86) | 56.6 (10.47)
Age, Customized [Number; unit: participants]
  <45 years | 46 | 33 | 46 | 125
  Between 45 to 64 years | 235 | 241 | 234 | 710
  ≥65 years | 74 | 78 | 84 | 236
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 151 | 159 | 442
  Male | 223 | 201 | 205 | 629
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 36 | 34 | 98
  Not Hispanic or Latino | 248 | 241 | 251 | 740
  Unknown or Not Reported | 79 | 75 | 79 | 233
Race (NIH/OMB) [Number; unit: participants] — A participant could have chosen more than 1 category for race; if so, they were included in each category indicated and were also included in the multiracial category.
  participants
    American Indian or Alaska Native | 2 | 5 | 5 | 12
    Asian | 13 | 11 | 11 | 35
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 3
    Black or African American | 80 | 80 | 80 | 240
    White | 261 | 258 | 267 | 786
    More than one race | 1 | 2 | 1 | 4
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 276 | 277 | 285 | 838
  Canada | 79 | 75 | 79 | 233
Weight [Mean (Standard Deviation); unit: kg] | 92.34 (20.296) | 91.47 (20.987) | 90.83 (18.590) | 91.54 (19.960)
Height [Mean (Standard Deviation); unit: cm] | 171.2 (10.15) | 169.3 (10.88) | 169.4 (10.15) | 170.0 (10.42)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.4 (5.94) | 31.9 (6.59) | 31.6 (5.92) | 31.6 (6.15)
Estimated glomerular filtration rate (eGFR) [Number; unit: participants] — eGFR based on calculated creatinine clearance.
  Categories:
  Normal renal function (≥90 mL/min/1.73 m2); Mild renal impairment(60 to <90 mL/min/1.73 m2); Moderate renal impairment (30 to <60 mL/min/1.73 m2) Severe renal impairment (0 to <30 mL/min/1.73 m2)
  participants
    ≥0 to <30 | 0 | 0 | 1 | 1
    ≥30 to <60 | 26 | 29 | 25 | 80
    ≥60 to <90 | 224 | 220 | 246 | 690
    ≥90 | 105 | 103 | 91 | 299
    Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough, Sitting, Clinic Systolic Blood Pressure.
Description: The change in sitting trough clinic systolic blood pressure measured at week 12 or final visit relative to baseline. Trough blood pressure is the average of the non-missing values of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 12.
Population: Full analysis set, all participants that took at least 1 dose of double-blind study drug and have a baseline and post-baseline value, with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 344 | 330 | 354
mmHg | -42.5 (0.81) | -44.0 (0.83) | -37.1 (0.80)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; Analysis of covariance (ANCOVA) model with treatment group as a fixed effect and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Overall Type 1 error rate of 0.05 controlled using 'Closed Testing' principle (hypothesis of "all treatment groups equal" first tested at 0.05 significance level; upon rejection of this hypothesis, pairwise comparison was tested at the 0.05 level; Mean Difference (Final Values) = -5.3, 95% CI [-7.6 to -3.1]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-9.2 to -4.6]

2. Secondary Outcome: Change From Baseline in Trough, Sitting, Clinic Systolic Blood Pressure.
Description: The change in sitting trough clinic systolic blood pressure measured at each week indicated relative to baseline. Trough blood pressure is the average of the non-missing values of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 355 | 352 | 364
mmHg
  Week 4 (n=343; n=330; n=352) | -34.7 (0.77) | -36.7 (0.79) | -29.7 (0.76)
  Week 8 (n=344; n=330; n=353) | -39.1 (0.78) | -39.4 (0.80) | -33.5 (0.77)

3. Secondary Outcome: Change From Baseline in Trough, Sitting, Clinic Diastolic Blood Pressure.
Description: The change in sitting trough clinic diastolic blood pressure measured at each week indicated relative to baseline. Trough blood pressure is the average (arithmetic mean) of the non-missing values of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline, Week 4, Week 8 and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 355 | 352 | 364
mmHg
  Week 4 (n=343; n=330; n=352) | -14.9 (0.46) | -15.8 (0.47) | -11.7 (0.45)
  Week 8 (n=344; n=330; n=353) | -17.0 (0.48) | -17.7 (0.49) | -13.9 (0.48)
  Week 12 (n=344; n=330; n=354) | -18.8 (0.47) | -20.5 (0.48) | -16.4 (0.46)

4. Secondary Outcome: Change From Baseline in Mean Trough Systolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in trough systolic blood pressure measured at week 12 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -32.9 (0.86) | -34.9 (0.90) | -25.9 (0.85)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at the 0.05 significance level; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-9.4 to -4.7]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at the 0.05 significance level; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-11.5 to -6.6]

5. Secondary Outcome: Change From Baseline in Mean Trough Diastolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in trough diastolic blood pressure measured at week 12 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -19.8 (0.55) | -20.2 (0.57) | -16.0 (0.54)

6. Secondary Outcome: Change From Baseline in 24-hour Mean Systolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -33.9 (0.76) | -36.3 (0.79) | -27.5 (0.75)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at the 0.05 significance level; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-8.5 to -4.3]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment group as a fixed effect and baseline value as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at the 0.05 significance level; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-11.0 to -6.7]

7. Secondary Outcome: Change From Baseline in 24-hour Mean Diastolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -19.4 (0.45) | -20.7 (0.46) | -16.2 (0.44)

8. Secondary Outcome: Change From Baseline in Mean Daytime (6 AM to 10 PM) Systolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 AM (inclusive) and 10 PM (exclusive).
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -35.3 (0.80) | -37.9 (0.84) | -28.8 (0.79)

9. Secondary Outcome: Change From Baseline in Mean Daytime (6 AM to 10 PM) Diastolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 AM (inclusive) and 10 PM (exclusive).
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -20.1 (0.48) | -21.8 (0.50) | -17.0 (0.47)

10. Secondary Outcome: Change From Baseline in Mean Nighttime (12 AM to 6 AM) Systolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in the mean nighttime (12am to 6am) systolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Mean nighttime is the average (arithmetic mean) of measurements recorded between the hours of 12 AM (inclusive) and 6 AM (exclusive).
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -29.6 (0.78) | -31.8 (0.81) | -23.9 (0.77)

11. Secondary Outcome: Change From Baseline in Mean Nighttime (12 AM to 6 AM) Diastolic Blood Pressure by Ambulatory Blood Pressure Monitoring.
Description: The change in the mean nighttime (12am to 6am) diastolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Mean nighttime is the average (arithmetic mean) of measurements recorded between the hours of 12 AM (inclusive) and 6 AM (exclusive).
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -17.5 (0.48) | -18.0 (0.50) | -14.0 (0.48)

12. Secondary Outcome: Change From Baseline in the Mean Systolic Blood Pressure at 0 to 12 Hours After Dosing by Ambulatory Blood Pressure Monitoring.
Description: The change in the mean 12 hour systolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The mean consists of the average (arithmetic mean) of measurements.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -36.2 (0.86) | -38.8 (0.89) | -29.7 (0.85)

13. Secondary Outcome: Change From Baseline in the Mean Diastolic Blood Pressure at 0 to 12 Hours After Dosing by Ambulatory Blood Pressure Monitoring.
Description: The change in the mean 12 hour diastolic blood pressure measured at week 12 or final visit relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The mean consists of the average (arithmetic mean) of measurements.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 232 | 214 | 238
mmHg | -20.4 (0.51) | -22.2 (0.53) | -17.5 (0.50)

14. Secondary Outcome: Change From Baseline in the Mean Systolic Blood Pressure During Each Hour of the 24-hour Ambulatory Blood Pressure Monitoring.
Description: The change from baseline for each hour interval of the 24-hour ambulatory blood pressure monitoring measured at week 12 or final visit. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The mean consists of the average (arithmetic mean) of measurements collected at each hour.
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 355 | 352 | 364
mmHg
  0 to 1 Hour (n=232; n=212; n=237) | -33.6 (0.96) | -36.2 (1.00) | -26.8 (0.95)
  1 to 2 Hour (n=232; n=214; n=238) | -33.4 (0.98) | -36.4 (1.02) | -27.5 (0.97)
  2 to 3 Hour (n=232; n=214; n=238) | -36.7 (1.02) | -39.3 (1.06) | -30.0 (1.00)
  3 to 4 Hour (n=232; n=214; n=238) | -36.6 (1.07) | -40.3 (1.12) | -29.6 (1.06)
  4 to 5 Hour (n=232; n=214; n=238) | -36.8 (1.07) | -40.8 (1.11) | -30.1 (1.06)
  5 to 6 Hour (n=232; n=214; n=238) | -37.2 (1.02) | -41.2 (1.06) | -31.5 (1.00)
  6 to 7 Hour (n=232; n=214; n=238) | -36.3 (1.04) | -38.6 (1.08) | -29.8 (1.02)
  7 to 8 Hour (n=232; n=214; n=238) | -37.2 (1.02) | -38.5 (1.06) | -29.7 (1.00)
  8 to 9 Hour (n=232; n=214; n=238) | -37.3 (1.02) | -38.1 (1.06) | -30.5 (1.01)
  9 to 10 Hour (n=232; n=214; n=238) | -36.9 (0.99) | -38.0 (1.04) | -30.8 (0.98)
  10 to 11 Hour (n=232; n=214; n=238) | -36.1 (1.02) | -37.6 (1.06) | -29.4 (1.01)
  11 to 12 Hour (n=232; n=214; n=238) | -35.2 (1.01) | -38.2 (1.05) | -29.3 (1.00)
  12 to 13 Hour (n=232; n=214; n=238) | -34.8 (1.05) | -36.2 (1.09) | -27.7 (1.04)
  13 to 14 Hour (n=232; n=214; n=238) | -34.1 (1.06) | -35.3 (1.11) | -26.4 (1.05)
  14 to 15 Hour (n=232; n=214; n=238) | -33.4 (1.06) | -35.0 (1.10) | -26.2 (1.04)
  15 to 16 Hour (n=232; n=214; n=238) | -30.9 (0.99) | -32.9 (1.03) | -25.3 (0.97)
  16 to 17 Hour (n=232; n=214; n=238) | -29.6 (0.94) | -31.1 (0.98) | -24.5 (0.93)
  17 to 18 Hour (n=231; n=214; n=238) | -28.5 (0.93) | -30.8 (0.97) | -23.1 (0.92)
  18 to 19 Hour (n=232; n=214; n=238) | -29.5 (0.90) | -31.9 (0.94) | -24.3 (0.89)
  19 to 20 Hour (n=232; n=214; n=238) | -29.7 (0.89) | -32.5 (0.93) | -23.5 (0.88)
  20 to 21 Hour (n=232; n=214; n=238) | -28.2 (0.94) | -31.2 (0.98) | -23.0 (0.92)
  21 to 22 Hour (n=232; n=214; n=238) | -30.6 (0.95) | -32.8 (0.99) | -24.6 (0.93)
  22 to 23 Hour (n=232; n=214; n=238) | -32.9 (0.94) | -34.0 (0.98) | -25.9 (0.92)
  23 to 24 Hour (n=232; n=214; n=238) | -33.1 (0.92) | -35.8 (0.96) | -26.1 (0.91)

15. Secondary Outcome: Change From Baseline in the Mean Diastolic Blood Pressure During Each Hour of the 24-hour Ambulatory Blood Pressure Monitoring.
Description: as for outcome 14
Time Frame: Baseline and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 355 | 352 | 364
mmHg
  0 to 1 Hour (n=232; n=212; n=237) | -18.2 (0.59) | -20.4 (0.62) | -15.2 (0.59)
  1 to 2 Hour (n=232; n=214; n=238) | -18.8 (0.65) | -20.9 (0.67) | -15.9 (0.64)
  2 to 3 Hour (n=232; n=214; n=238) | -21.2 (0.66) | -23.4 (0.69) | -17.7 (0.65)
  3 to 4 Hour (n=232; n=214; n=238) | -20.8 (0.69) | -23.7 (0.72) | -18.2 (0.68)
  4 to 5 Hour (n=232; n=214; n=238) | -21.7 (0.67) | -23.7 (0.70) | -17.9 (0.66)
  5 to 6 Hour (n=232; n=214; n=238) | -20.9 (0.67) | -23.6 (0.70) | -19.0 (0.66)
  6 to 7 Hour (n=232; n=214; n=238) | -20.8 (0.65) | -22.0 (0.67) | -18.0 (0.64)
  7 to 8 Hour (n=232; n=214; n=238) | -20.5 (0.66) | -21.9 (0.69) | -17.7 (0.65)
  8 to 9 Hour (n=232; n=214; n=238) | -20.7 (0.67) | -21.5 (0.69) | -17.9 (0.66)
  9 to 10 Hour (n=232; n=214; n=238) | -21.0 (0.66) | -21.9 (0.68) | -18.3 (0.65)
  10 to 11 Hour (n=232; n=214; n=238) | -19.7 (0.67) | -20.7 (0.70) | -16.7 (0.66)
  11 to 12 Hour (n=232; n=214; n=238) | -19.3 (0.69) | -21.2 (0.72) | -17.0 (0.68)
  12 to 13 Hour (n=232; n=214; n=238) | -19.2 (0.73) | -20.3 (0.76) | -16.0 (0.72)
  13 to 14 Hour (n=232; n=214; n=238) | -19.6 (0.72) | -19.5 (0.75) | -15.3 (0.71)
  14 to 15 Hour (n=232; n=214; n=238) | -18.9 (0.72) | -19.7 (0.75) | -15.4 (0.71)
  15 to 16 Hour (n=232; n=214; n=238) | -17.8 (0.65) | -18.6 (0.68) | -14.5 (0.65)
  16 to 17 Hour (n=232; n=214; n=238) | -17.2 (0.65) | -16.9 (0.68) | -13.9 (0.64)
  17 to 18 Hour (n=231; n=214; n=238) | -16.6 (0.64) | -17.1 (0.66) | -13.2 (0.63)
  18 to 19 Hour (n=232; n=214; n=238) | -17.4 (0.65) | -18.1 (0.67) | -14.3 (0.64)
  19 to 20 Hour (n=232; n=214; n=238) | -17.8 (0.60) | -18.5 (0.63) | -13.8 (0.60)
  20 to 21 Hour (n=232; n=214; n=238) | -16.7 (0.64) | -18.4 (0.67) | -13.9 (0.63)
  21 to 22 Hour (n=232; n=214; n=238) | -17.8 (0.66) | -18.5 (0.69) | -14.7 (0.65)
  22 to 23 Hour (n=232; n=214; n=238) | -19.5 (0.62) | -19.6 (0.65) | -15.6 (0.62)
  23 to 24 Hour (n=232; n=214; n=238) | -20.2 (0.60) | -21.0 (0.62) | -16.4 (0.59)

16. Secondary Outcome: Percentage of Participants Who Reached Target Clinic Systolic Blood Pressure of <140 mm Hg and/or Reduction of ≥20 mm Hg From Baseline.
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at each week indicated, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the arithmetic mean of the non-missing values of the 3serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline, Week 4, Week 8 and Week 12.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 355 | 352 | 364
percentage of participants
  Week 4 (n=343; n=330; n=352) | 87.8 | 90.0 | 79.8
  Week 8 (n=344; n=330; n=353) | 93.3 | 92.4 | 85.6
  Week 12 (n=344; n=330; n=354) | 93.0 | 94.2 | 89.3

17. Secondary Outcome: Percentage of Participants Who Reached Target Clinic Diastolic Blood Pressure of <90 mm Hg and/or Reduction of ≥10 mm Hg From Baseline.
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at each week indicated, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the arithmetic mean of the non-missing values of the 3 serial trough sitting diastolic blood pressure measurements.
Time Frame: Baseline, Week 4, Week 8 and Week 12.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 355 | 352 | 364
percentage of participants
  Week 4 (n=343; n=330; n=352) | 89.2 | 89.7 | 85.2
  Week 8 (n=344; n=330; n=353) | 90.7 | 90.9 | 87.8
  Week 12 (n=344; n=330; n=354) | 94.5 | 95.8 | 91.5

18. Secondary Outcome: Percent of Participants Who Reached Target Clinic Systolic Blood Pressure of <140 mm Hg and/or Reduction of ≥20 mm Hg From Baseline and Target Clinic Diastolic Blood Pressure of <90 mm Hg and/or Reduction of ≥10 mm Hg From Baseline.
Description: Percentage of participants who achieve both a clinic diastolic and systolic blood pressure response measured at each week indicated, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg AND less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Diastolic and systolic blood pressure is based on the arithmetic mean of the non-missing values of the 3 serial trough sitting blood pressure measurements.
Time Frame: Baseline, Week 4, Week 8 and Week 12.
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 355 | 352 | 364
percent of participants
  Week 4 (n=343; n=330; n=352) | 81.3 | 84.8 | 74.4
  Week 8 (n=344; n=330; n=353) | 88.1 | 87.3 | 81.0
  Week 12 (n=344; n=330; n=354) | 91.3 | 92.4 | 84.7

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Serious Adverse Events (participants affected / at risk) | 1/355 | 10/352 | 8/364
Other Adverse Events (participants affected / at risk) | 141/355 | 144/352 | 94/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD (N=355) | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD (N=352) | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD (N=364)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0
Accelerated hypertension (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20-40mg/Chlorthalidone 12.5-25mg QD (N=355) | Azilsartan Medoxomil 40-80mg/Chlorthalidone 12.5-25mg QD (N=352) | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD (N=364)
Fatigue (General disorders) | 33 | 14 | 16
Blood creatinine increased (Investigations) | 66 | 78 | 34
Blood uric acid increased (Investigations) | 19 | 17 | 12
Dizziness (Nervous system disorders) | 41 | 58 | 29
Headache (Nervous system disorders) | 19 | 13 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.